CLINICAL TRIAL: NCT06686576
Title: A Phase Ib/III, Open-Label, Randomized Study of Neoadjuvant QL1706 Versus Standard of Care in Participants With Untreated of Microsatellite Instability-high or Mismatch Repair-deficient, Resectable Colon Cancer
Brief Title: A Study of Neoadjuvant QL1706 in Participants With Untreated dMMR/MSI-H Resectable Colon Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QL1706-307
Record Dates: First submitted 2024-11-11; First posted 2024-11-13 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Phase Ib/Ⅲ Participants will receive QL1706 pre surgery
  Interventions: Drug: QL1706
- Phase III Control group (Active Comparator): Participants will receive SOC (CAPEOX/Capecitabine) or undergo expectant observation post surgery.
  Interventions: Drug: CAPEOX/Capecitabine

INTERVENTIONS:
Drug: QL1706 — Phase Ib/Ⅲ： QL1706 will be administered
  Arms: Experimental group
Drug: CAPEOX/Capecitabine — Phase Ⅲ：CAPEOX/Capecitabine will be administered
  Arms: Phase III Control group

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of neoadjuvant QL1706 in participants with untreated T4N0 or Stage III (resectable), microsatellite instability high/ defective mismatch repair (MSI-H/dMMR) colon cancer

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent;
* Eastern Cooperative Oncology Group Performance Status of 0 or 1
* Untreated pathologically confirmed colon adenocarcinoma
* Radiographic assessment showed a resectable stage IIB-III based on AJCC Stage VIII (cT4 or cN+ only).
* Has a tumor demonstrating the presence of MSI-H/ dMMR
* Adequate organ function as described in the protocol

Exclusion Criteria:

* Previously received any antitumor therapy for the disease under study, including surgery, radiotherapy, chemotherapy, targeted therapy, immunotherapy, etc
* Has distant metastatic disease.
* Has an active autoimmune disease that has required systemic treatment in past 2 years
* Has know history of, or any evidence of interstitial lung disease;
* Has an active infection requiring systemic therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 363 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response(pCR), defined as the proportion of subjects with no residual tumor in the primary tumor removed and in all lymph nodes removed after neoadjuvant therapy. | 1 month after surgery
Event Free Survival, EFS(EFS), defined as the time from randomization to either disease recurrence or death due to any cause or treatment related toxicity that results in the participant not being suitable for surgery. | Up to approximately 5 years

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to approximately 5 years
  OS is defined as time from randomization to death from any cause
R0 tumor resection rate | 2 week after surgery
  R0 tumor resection rate is defined as the proportion of subjects with R0 excision
Number of Participants with treatment emergent adverse events (AEs), serious adverse events (SAEs), Immune-mediated Adverse Event (imAEs), AEs leading to death and AEs leading to discontinuation of study treatment | Up to approximately 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Cancer Hospital of Sun Yat-sen University, Guangzhou, China